CLINICAL TRIAL: NCT04205825
Title: Development and Evaluation of the Impact of a Safety Checklist Adapted to Interventional Cardiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IIBSP-LVS-2017-49
Record Dates: First submitted 2019-12-12; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Complication of Surgical Procedure
Keywords: Nursing; Patient Safety; Checklist; Cardiology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Safety Checklist (Experimental): Patients randomized in the New Safety Checklist intervention, nurses will use the New Safety Checklist, which we have named: INCARDIO-PASS (Interventional CARDIOlogy-Patient Safety System) checklist.
  Interventions: Other: The New Safety Checklist
- Habitual Practice (No Intervention): Patients randomized in this arm they will receive the habitual practice.

INTERVENTIONS:
Other: The New Safety Checklist — Patients randomized in the New Safety Checklist intervention, nurses will use the New Safety Checklist, which we have named: INCARDIO-PASS (Interventional CARDIOlogy-Patient Safety System) checklist.
  Arms: New Safety Checklist

SUMMARY:
The hypothesis is that patients undergoing cardiac catheterization, in which the New Safety Checklist has been used, have fewer perioperative complications compared to patients in which the habitual practice has been used.

DETAILED DESCRIPTION:
The aim of this study is to develop a New Safety Checklist in perioperative patients undergoing cardiac catheterization in interventional cardiology units and assess it impact on the incidence of perioperative complications compared to habitual practice.

The study will consist in two phases; the first phase: development of the New Safety Checklist, and the second phase will be a multicenter randomized clinical trial, a parallel two-arm corresponding to the use of the New Safety Checklist compared to the habitual practice in all patients undergoing cardiac catheterization in interventional cardiology units, according to the inclusion criteria..

The expected number of patients in this trial will be 6000. The principal outcome of this study will be: the incidence of perioperative complications. The secondary outcomes will be: socio-demographic data, clinical patient data and procedure type data. Data collection will be done through reviewing clinical history.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) undergoing cardiological intervention in hemodynamic units and interventionist cardiology.
* Patients who accept to participate in the study.

Exclusion Criteria:

* Patients undergoing urgent procedure.
* Patients requiring ventilatory support or in a situation of hemodynamic instability.
* Patients with cognitive impairment, mental disability or other serious difficulty in communication.
* Patients with insufficient fluidity of the main languages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
INCIDENCE of PERIOPERATIVE COMPLICATIONS | from the discharge or up to 24 hours post-procedure
  The perioperative complications will be collected after randomization, from discharge or up to24 hours post-procedure.
  The clinical history will be reviewed to evaluate the incidence of complications. Expected complications will be: severe systemic complications (major cardiovascular events [MACE], coronary artery complications, and structural complications), peripheral vascular complications, and reactions to contrast media.

SECONDARY OUTCOMES:
Socio-demographic data | from the discharge or up to 24 hours post-procedure
  Socio-demographic data will be collected after randomization, from the discharge or up to 24 hours post-procedure.
  The clinical history will be reviewed to collect socio-demographic data: gender (male/female), age (absolute value), weight (kilograms) and height (centimeters).
Clinical data | from the discharge or up to 24 hours post-procedure
  Clinical data will be collected after randomization, from the discharge or up to 24 hours post-procedure.
  The clinical history will be reviewed to collect cardiovascular risk factors (dyslipemia, smoking), clinical record (medical allergies, ischemic, valvular heart disease, cardiomyopathy, arrhythmias, disease pulmonary, platelet antiaggregant treatment).
Procedure data | from the discharge or up to 24 hours post-procedure
  Procedure data will be collected after randomization, from the discharge or up to 24 hours post-procedure.
  The clinical history will be reviewed to collect procedure data, tipe of procedure done (coronary, structural, diagnostic procedure, right catheterization).

CONTACTS AND LOCATIONS:
Locations (1):
- FGS Hospital de la Santa Creu i Sant Pau, Barcelona, Spain